CLINICAL TRIAL: NCT06996743
Title: Effect of Pilates Exercises on Menopausal Symptoms in Postmenopausal Obesity
Brief Title: Effect of Pilates Exercises on Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, merve yiğit kocamer, lecturer, Batman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BU-FTR-MYK-01
Record Dates: First submitted 2025-05-07; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Menopausal; Obese Patients; Pilates Exercise; Quality of Life and Menopause
Keywords: menopause; obese women; pilates exercises; blood lipid profile

STUDY DESIGN:
Intervention Model Description: 1. Reformer pilates group
  2. Mat pilates group
  3. Lifestyle change group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- reformer pilates group (Active Comparator): It was done by a specialist physiotherapist on a Pilates reformer device, and the exercises lasted approximately 60 minutes. The exercise content consists of strengthening exercises, stretching exercises, and warm-up and cool-down exercises.
  The program was updated with the addition of a new exercise type every two weeks.
  The repetition numbers were updated to 8 repetitions in the first two weeks, 10 repetitions in the third and fourth weeks, and 12 repetitions in the last four weeks.
  Interventions: Other: reformer pilates group
- 2- Mat pilates group (Active Comparator): The special exercises in the reformer pilates program were applied as structured mat pilates. First, the exercises to be done by the physiotherapist were taught. Then, an illustrated brochure with the exercises was prepared by the expert physiotherapist and distributed to the participants in this group. In order for the exercise to be done correctly and effectively, a video shot by the expert physiotherapist was sent to the patients in addition to the brochure. Each exercise was explained in detail in the video and the tricks were mentioned. The patient did the exercises at home. Online control was provided via smartphone once a week and the exercises were done under the observation of the expert physiotherapist during the online interview. The exercise follow-up chart was filled out regularly twice every week. The exercise duration lasted approximately 60 minutes. The program was updated with the addition of a new exercise type every two weeks and continued in its fixed form for the
  Interventions: Other: Mat pilates group
- 3- Lifestyle change group (Active Comparator): After the doctor's check-up, routine application continued. The patient was informed about physical activity. In addition; a physical activity-based brochure prepared by the Specialist Physiotherapist was distributed to the participants in this group. The brochure included methods for coping with menopause and lifestyle changes to reduce symptoms.
  Interventions: Other: Lifestyle change group

INTERVENTIONS:
Other: reformer pilates group — Reformer Pilates exercises were applied to the pilates group twice a week for a total of 8 weeks.
  Arms: reformer pilates group
Other: Mat pilates group — Mat Pilates exercises were applied to the pilates group twice a week for a total of 8 weeks.
  Arms: 2- Mat pilates group
Other: Lifestyle change group — After the doctor's check-up, routine application continued. The patient was informed about physical activity. In addition; a physical activity-based brochure prepared by the Specialist Physiotherapist was distributed to the participants in this group.
  Arms: 3- Lifestyle change group

SUMMARY:
Menopause, a significant transition in a woman's life characterized by the cessation of menstruation and a decline in ovarian function, leads to reduced levels of estrogen and progesterone. This hormonal shift is associated with a range of symptoms that can adversely affect women's quality of life, including vasomotor symptoms such as hot flashes and night sweats, psychological symptoms like mood swings and depression, as well as urogenital symptoms such as vaginal dryness and sexual dysfunction. These symptoms, collectively referred to as menopausal symptoms, can vary in severity and duration and frequently require intervention to alleviate their impact on daily life.

DETAILED DESCRIPTION:
The aim of our study was to determine the effect of pilates exercises on menopausal symptoms in postmenopausal obesity and to compare it with the control group. The study was designed as a single-blind randomized controlled trial. 45 obese individuals in the postmenopausal period were included in the study. The patients were randomly divided into 3 groups and a total of 16 treatment sessions were applied to both groups for 8 weeks, 2 days a week. No exercise intervention was applied to the control group. Reformer Pilates exercises were applied to Group 1, and mat Pilates exercises were applied to Group 2. A physical activity-based brochure including lifestyle changes was distributed to Group 3. A total of two evaluations were made before and after exercise. In the evaluation, the Menopausal Symptoms RatingScale (MRS) for menopausal symptoms, the Menopause-Specific Quality of Life Assessment Scale (MENQOL) for quality of life assessment, the Beck Depression Inventory (BDI) for depression, the Pittsburgh Sleep Quality Index (PSQI) for assessing sleep quality, the Six-Minute Walking Test (6 MWT) for assessing aerobic capacity, the Body Analysis Scale (TANITA) for assessing body composition, and laboratory analyses of blood samples taken for assessing blood lipid profile were used. Statistical analyses were performed to compare the data.

ELIGIBILITY:
Inclusion Criteria:

* Women who have entered menopause
* Being diagnosed with obesity (30 kg/m2 ≤ BMI ≤ 40 kg/m2 )
* Having the physical or cognitive ability to exercise
* Being sedentary ('International Physical Activity Questionnaire' will be used. Those in the Inactive Category group will be included.)
* Those who agree to participate in the study

Exclusion Criteria:

* BMI below 30
* Those with serious heart disease, DM, kidney, liver, thyroid disease and cancer
* Those receiving hormone therapy
* Those using antipsychotic drugs
* Those using steroids and derivatives
* Those using insulin-sensitizing drugs
* Those with musculoskeletal diseases that will prevent exercise • Cognitive problems that will affect cooperation

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — FEMALE
Enrollment: 45 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Menopause Symptoms Assessment Scale (MSAS) | 8 week
  The Menopause Symptoms Assessment Scale (MSS) is a very useful tool for assessing the symptoms of women in menopause and measuring their impact on their quality of life. Using a Likert-type scale, determining the severity of symptoms provides important data for treatment and intervention planning.
  In particular, being organized in 3 sub-dimensions (somatic, psychological and urogenital complaints) helps understand the different aspects of menopause. This diversity provides a comprehensive assessment for both health professionals and researchers. The Likert-type scale, which includes menopausal complaints, is scored between 0 and 4. It indicates that the complaint is not present at all, while 4 indicates that it is very severe. The total score of the scale is calculated with the scores obtained from each item.high score indicates negativity
Menopause-Specific Quality of Life Scale (MSQLS) | 8 week
  The Menopause-Specific Quality of Life Scale (MSQLS) is a comprehensive tool that multi-dimensionally assesses the quality of life of women in the menopausal process. Developed by Hilditch and colleagues, this scale focuses on the physical, psychosocial, sexual and vasomotor symptoms of menopause, revealing the impact of different symptoms on quality of life in more detail.
  Especially the Likert-type assessment consisting of 32 questions and scored from 1 to 8 is very useful in examining the severity of problems in the menopausal process. Such a scale is an important tool for understanding the difficulties experienced by women in the menopausal period and for making appropriate interventions. The scoring of each subdomain helps determine the degree to which problems specific to that subject cause discomfort, which allows for more effective development of treatment and support plans. The lowest score is 8 and the highest score is 256. High score indicates negativity

SECONDARY OUTCOMES:
Beck Depression Inventory | 8 week
  The Beck Depression Inventory (BDI) is a tool that can effectively assess the severity of depression and changes in an individual's mood. Developed in 1961 by Aaron T. Beck and his colleagues, it specifically measures how individuals feel, focusing on the cognitive and emotional dimensions of depression.
  There are 21 questions in total, the item is scored between 0-3 and provides information about different levels of depression. The BDI, which is measured with a minimum score of 0 and a maximum score of 63 points, is a highly functional method for determining the severity of depression. A high score indicates increased violence, which is a negative situation.
Pittsburgh Sleep Quality Index (PSQI) | 8 week
  The Pittsburgh Sleep Quality Index (PSQI) is an effective scale with a wide scope for assessing sleep quality. Developed in 1989 by Buysse and colleagues, this scale consists of a series of questions aimed at understanding various dimensions of sleep and offers a multifaceted approach to more accurately assess sleep disorders. This scale evaluates an individual's sleep according to various factors (e.g., sleep duration, time to fall asleep, and difficulty felt upon waking).
  This scale, consisting of 24 questions, consists of 19 questions based on the individual's self-assessment and 5 questions answered by the spouse or roommate. Such a structure evaluates the individual's sleep quality from a broader perspective, taking into account the effects of possible . A high score indicates increased violence, which is a negative situation.
Body Composition | 8 week
  Measurement was made with Tanita body analysis scale. (TANITA TT 730 MA)
  The height and weight of the patients were measured by the same person with standardized devices. Body mass index (BMI) is obtained by dividing the body weight measured in kilograms by the square of the height in meters. This method is a practical classification tool widely used to determine whether the individual is underweight, normal weight, overweight or obese. Waist circumference measurement was made with a tape measure at the level of the navel, with the individuals in an upright position and the abdomen relaxed. During the measurement, the tape measure was used in a way that it would touch the skin without applying pressure.
BLOOD LIPID PROFILE | 8 week
  During routine doctor visits, patients' blood values are routinely checked by the hospital's specialist doctor. The blood values already taken/taken will be used.
  Total cholesterol (TC)
  High-density lipoprotein (HDL)
  Low-density lipoprotein (LDL)
  Triglyceride (TG)
AEROBIC CAPACITY | 8 week
  The Six Minute Walk Test (6MWT) is a practical, reliable and widely used measurement method for evaluating an individual's cardiopulmonary functions and general physical endurance level. This test is widely used especially in the evaluation of disorders in the respiratory or cardiovascular systems. The purpose of the test is to observe the individual's performance during physical exercise, to evaluate the level of fatigue and to determine the level of endurance. The use of the Modified Borg Scale in the assessment of dyspnea increases the reliability and validity of the test. The Borg scale is a common tool for measuring the severity of dyspnea and allows the patient to express their symptoms numerically. The 0-10 rating scale is a practical measurement tool that allows the patient to subjectively assess the severity of dyspnea they experience. In this system, "0" represents no dyspnea, while "10" represents the most severe and intolerable dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Merve YİĞİT KOCAMER MERVE, Principal Investigator — Batman University
Locations (2):
- Turkey (Türkiye) (2):
  - Batman Center, Batman, Gültepe
  - Batman, Batman

IPD SHARING:
Plan to Share IPD: No